CLINICAL TRIAL: NCT06001905
Title: Research on the Construction of Cord Blood Storage Decision Aid Network Platform Based on "Internet +"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Shandong Nursing Association (Unknown)
Responsible Party: Principal Investigator, Hong Ji, chief superintendent nurse, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2023(059)
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Pregnant Women

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cord blood, as an important alternative source of hematopoietic stem cells, can be used to reconstruct bone marrow hematopoietic and immune function, and is an effective means to treat children with blood diseases. However, at present, the collection rate of cord blood is not high in our country, only the mother have the right to decide whether or not. At the same time, domestic studies on cord blood collection are still very limited, for the lack of effective programs and policies, which can not provide help to improve the collection level of cord blood. Therefore, in order to improve the rate of umbilical cord blood collection, it is particularly necessary to build tools to help pregnant women decide whether to retain cord blood. This topic will investigate and analyze the cognition and retention intention of pregnant women for umbilical cord blood collection. At the same time, the related process of pregnant women for umbilical cord blood retention will be deeply explored. Based on the results of quantitative and qualitative investigation, Internet technology will be used to build a network platform for pregnant women for umbilical cord blood storage decision AIDS, and the effectiveness of this tool will be evaluated. To provide theoretical basis for clinical medical workers and umbilical cord blood bank staff to establish the decision plan of cord blood storage.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old;

  * Pregnant women whose gestational age ≥12 weeks and registered in our hospital;

    * With a certain level of education, can complete the questionnaire independently;

      * Informed consent to participate in the study

Exclusion Criteria:

* There are patients with mental illness;

  * Participated in other clinical studies in the past three months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Only pregnant women have the right to decide whether to store umbilical cord blood. Therefore, pregnant women who have been registered in our hospital were selected in this study. The first test should be performed after 12 weeks of gestation, so pregnant women over 12 weeks of gestation should be selected.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Construct the network platform of cord blood storage decision aid tool | 2024.07.10
  Construct the network platform of cord blood storage decision aid tool based on "Internet +" and apply it to clinical practice to provide support and help for pregnant women in cord blood storage decision, avoid decision regret, and improve pregnant women's willingness and satisfaction in cord blood storage.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongguo, Jinan, China

IPD SHARING:
Plan to Share IPD: No